CLINICAL TRIAL: NCT04163484
Title: Contrast-associated Acute Kidney Injury in Patients With Different Types of Coronary Artery Disease
Status: Completed | Type: Observational
Sponsor: I.M. Sechenov First Moscow State Medical University (Other)
Responsible Party: Principal Investigator, Olga Mironova, MD PhD Associate Professor, I.M. Sechenov First Moscow State Medical University
Other Study IDs: 11/2019
Record Dates: First submitted 2019-10-25; First posted 2019-11-14 (Actual); Last update posted 2024-10-08 (Actual); Status verified 2024-10

CONDITIONS: Coronary Artery Disease; Angina, Unstable; Angina, Stable; STEMI - ST Elevation Myocardial Infarction; NSTEMI - Non-ST Segment Elevation MI; Contrast-induced Nephropathy; Acute Kidney Injury
Keywords: coronary artery disease; iodinated contrast media; stable angina; unstable angina; STEMI; NSTEMI; PCI; acute kidney injury
MeSH Terms: conditions — Coronary Artery Disease; Angina, Unstable; Angina, Stable; ST Elevation Myocardial Infarction; Non-ST Elevated Myocardial Infarction; Acute Kidney Injury

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Stable coronary artery disease
  Interventions: Other: Iodinated contrast
- ST-elevation myocardial infarction
  Interventions: Other: Iodinated contrast
- Non-ST-elevation myocardial infarction
  Interventions: Other: Iodinated contrast

INTERVENTIONS:
Other: Iodinated contrast — Intra-arterial injection of iodinated contrast media during percutaneous coronary intervention

SUMMARY:
The goal of the study is to assess the prevalence of contrast-associated acute kidney injury in patients with stable coronary artery disease, ST-elevation myocardial infarction and unstable angina/NSTEMI, assess the risk factors of contrast-induced acute kidney injury development and the influence of contrast-induced kidney injury on 1-year prognosis.

ELIGIBILITY:
Inclusion Criteria:

* Males and females aged 18-80
* Stable CAD receiving optimal medical treatment requiring PCI or STEMI or NSTEMI
* Intra-arterial injection of iodinated contrast media
* Informed consent

Exclusion Criteria:

* Age less than 18
* Pregnancy, lactation
* Refuse to sign the informed consent
* Contraindications for PCI
* Other conditions affecting prognosis (oncology, liver failure etc)
* CKD stage 4-5
* Patients receiving nephrotoxic drugs

Ages: 18 Years to 80 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Males and females aged 18-80, who have the indication for treatment of CAD with PCI requiring the intra-arterial injection of iodinated contrast-media
Sampling Method: Probability Sample
Enrollment: 156 (Actual)
Dates: Start 2019-01-15 (Actual); Primary Completion 2022-12-30 (Actual); Study Completion 2024-05-30 (Actual)

PRIMARY OUTCOMES:
Contrast associated acute kidney injury | 48-72 hours
  Number of patients with contrast associated kidney injury after contrast exposure

SECONDARY OUTCOMES:
Overall mortality | 1 year
Cardiovascular mortality | 1 year
Myocardial infarction | 1 year
  Number of patients with myocardial infarction
Stroke | 1 year
Repeat revascularization | 1 year
  PCI or CABG
Repeat hospitalisation | 1 year
Acute decompensation of heart failure | 1 year
  Number of patients with acute decompensation of heart failure
Chronic kidney disease progression | 1 year
  Progression of chronic kidney disease in patients with decreased glomerular filtration rate on inclusion
New-onset dialysis | 1 year
  Number of patients with new-onset dialysis

CONTACTS AND LOCATIONS:
Overall Officials: Olga Mironova, MD PhD, Study Director — I. M. Sechenov First Moscow State Medical University (Sechenov University)
Locations (1):
- Sechenov University, Moscow, Russia

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- See also: Kuznetsov VA, Mironova OIu, Gritsanchuk AM, Fomin VV. Contrast-associated acute kidney injury after percutaneous coronary interventions in patients with acute coronary syndrome: a real-world study. Consilium Medicum. 2022;24(10):713-717 — http://doi.org/10.26442/20751753.2022.10.201925